CLINICAL TRIAL: NCT05281302
Title: Innovative Therapy Combining Neck Muscle Vibration and Transcranial Direct Current Stimulation in Association With Conventional Rehabilitation in Left Unilateral Spatial Neglect Patients: HEMISTIM Protocol
Brief Title: Combination of Neck Muscle Vibration and tDCS With Conventional Rehabilitation in Neglect Patients
Acronym: HEMISTIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technological problem
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Collaborators: Université de Lorraine, DevAH (EA3450), Nancy, France (Unknown); Union de Gestion des Etablissements des Caisses d'Assurance Maladie - PACA (Unknown); Institut Régional de Médecine Physique et de Réadaptation de Nancy - Etablissement de Lay Saint Christophe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRR-LSC-2021-1
Record Dates: First submitted 2022-02-21; First posted 2022-03-16 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Unilateral Spatial Neglect
Keywords: Neck muscle vibration; tDCS; conventional rehabilitation; neglect

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control patients (No Intervention): Patient receiving no additional treatment to conventional occupational therapy sessions
- left-NMV (Experimental): Patient will be equipped with vibratory stimulators during conventional occupational therapy sessions.
  Only the left-side NMV vibrator will be activated.
  Interventions: Device: Neck muscle vibration
- left-NMV + sham-tDCS (Sham Comparator): Patient will be equipped with vibratory stimulators and with electrodes form sham-tDCS during conventional occupational therapy sessions.
  Only the left-side NMV vibrator will be activated.
  Interventions: Device: Neck muscle vibration + sham-tDCS
- left-NMV + anodal-tDCS (Experimental): Patient will be equipped with vibratory stimulators and with electrodes for tDCS during conventional occupational therapy sessions.
  Only the left-side NMV vibrator will be activated.
  Interventions: Device: Neck muscle vibration + anodal-tDCS

INTERVENTIONS:
Device: Neck muscle vibration — Patient will receive neck muscle vibration during the first 15 minutes of occupational therapy. Vibratory stimulators will be fixed bilaterally on the skin over the belly of the trapezius muscles and fastened with straps. Only the left vibrator will be activated.
  Arms: left-NMV
Device: Neck muscle vibration + sham-tDCS — Patient will receive neck muscle vibration during the first 15 minutes of occupational therapy.. Vibratory stimulators will be fixed bilaterally on the skin over the belly of the trapezius muscles and fastened with straps. Only the left vibrator will be activated.
  Moreover, tDCS will be applied using an electrical stimulator (DC-STIMULATOR®, NeuroCare, Illmenau, Germany) through large saline-soaked sponge surface electrodes placed as follows: anode over the right (ipsilesional) posterior parietal cortex (P4 according to the International 10-20 EEG electrode placement system) and cathode over the left supraorbital region. The tDCS will be automatically turned off after 20 seconds. This allows the reproduction of the initial mild itching sensation at the beginning of active tDCS, thus ensuring that the patient stays blind to the activation status of the device.
  Arms: left-NMV + sham-tDCS
Device: Neck muscle vibration + anodal-tDCS — Patient will receive neck muscle vibration during the first 15 minutes of occupational therapy. Vibratory stimulators will be fixed bilaterally on the skin over the belly of the trapezius muscles and fastened with straps. Only the left vibrator will be activated.
  Moreover, tDCS will be applied using an electrical stimulator (DC-STIMULATOR®, NeuroCare, Illmenau, Germany) through large saline-soaked sponge surface electrodes placed as follows: anode over the right (ipsilesional) posterior parietal cortex (P4 according to the International 10-20 EEG electrode placement system) and cathode over the left supraorbital region. A continuous 2 mA current will be delivered for 20 minutes simultaneously to NMV stimulation. The stimulation will begin 5 minutes before the beginning of occupational therapy.
  Arms: left-NMV + anodal-tDCS

SUMMARY:
BACKGROUND: Unilateral spatial neglect (USN) rehabilitation remains a challenge and requires the development of new methods that can be easily integrated into conventional practice. The aim of the HEMISTIM protocol is to assess immediate and long-term functional outcomes and neuropsychological aspects of recovery, induced by an innovative association of left-side neck-muscle vibration (NMV) and anodal transcranial Direct Current Stimulation (tDCS) on the ipsilesional posterior parietal cortex during occupational therapy sessions in patients with left USN.

METHODS: Participants will be randomly assigned to 4 groups: control, Left-NMV, Left-NMV + sham-tDCS or Left-NMV + anodal-tDCS. NMV will be applied during the first 15 minutes of occupational therapy and tDCS will be applied for 20 minutes, starting 5 minutes before, three days a week for three weeks. USN will be assessed at baseline, just at the end of the first experimental session, after the first and third weeks of the protocol and three weeks after its ending.

DISCUSSION: Left NMV, by activating multisensory integration neuronal networks, might enhance beneficial effects obtained by conventional occupational therapy sessions since interesting post-effects were shown when it was combined with voluntary upper limb movements. The investigators expect to reinforce lasting intermodal recalibration through LTP-like plasticity induced by anodal tDCS. The HEMISTIM protocol represents a therapeutic innovation associated to conventional practice that could provide a partial solution to the rehabilitation challenges of the USN syndrome and some insights to its underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* admitted in a post-stroke rehabilitation unit in the sub-acute phase (15 days to 6 months from the onset of stroke symptoms)
* at least 18 years old
* a first unilateral right hemispheric stroke
* diagnosis of stroke confirmed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Behavioral Inattention Test (c-BIT), inferior or equal to 129

Exclusion Criteria:

* unable to give informed consent
* pregnant women
* patients with skin lesions on the areas for electrode placement
* having history of metal-in-cranial injury
* epilepsy
* vestibulo-cochlear illness
* cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Catherine Bergego Scale | at the end of the first week of inclusion
  Functional scale assessing unilateral spatial neglect severity in daily life situations. This is a score on 30. The higher the score, the severe the unilateral spatial neglect
Catherine Bergego Scale | Immediately following first session of occupational therapy.
  Functional scale assessing unilateral spatial neglect severity in daily life situations. This is a score on 30. The higher the score, the severe the unilateral spatial neglect
Catherine Bergego Scale | after the first week of protocol
  Functional scale assessing unilateral spatial neglect severity in daily life situations. This is a score on 30. The higher the score, the severe the unilateral spatial neglect
Catherine Bergego Scale | after the third week of protocol
  Functional scale assessing unilateral spatial neglect severity in daily life situations. This is a score on 30. The higher the score, the severe the unilateral spatial neglect
Catherine Bergego Scale | 3 weeks after the last session of intervention
  Functional scale assessing unilateral spatial neglect severity in daily life situations. This is a score on 30. The higher the score, the severe the unilateral spatial neglect

SECONDARY OUTCOMES:
Fluff test | at the end of the first week of inclusion
  Investigating personal neglect with targets sticked on patients' clothes. The number of targets removed targets will be counted in order to calculate a score of personal neglect expressed as the difference of percentages of targets found on each side of the body (left-right), this value becoming more negative with the severity of personal neglect.
Fluff test | Immediately following first session of occupational therapy.
  Investigating personal neglect with targets sticked on patients' clothes. The number of targets removed targets will be counted in order to calculate a score of personal neglect expressed as the difference of percentages of targets found on each side of the body (left-right), this value becoming more negative with the severity of personal neglect.
Fluff test | after the first week of protocol
  Investigating personal neglect with targets sticked on patients' clothes. The number of targets removed targets will be counted in order to calculate a score of personal neglect expressed as the difference of percentages of targets found on each side of the body (left-right), this value becoming more negative with the severity of personal neglect.
Fluff test | after the third week of protocol
  Investigating personal neglect with targets sticked on patients' clothes. The number of targets removed targets will be counted in order to calculate a score of personal neglect expressed as the difference of percentages of targets found on each side of the body (left-right), this value becoming more negative with the severity of personal neglect.
Fluff test | 3 weeks after the last session of intervention
  Investigating personal neglect with targets sticked on patients' clothes. The number of targets removed targets will be counted in order to calculate a score of personal neglect expressed as the difference of percentages of targets found on each side of the body (left-right), this value becoming more negative with the severity of personal neglect.
Gainotti's drawing copying test | at the end of the first week of inclusion
  Informs us on two kinds of peri-personal neglect referring to distinct disturbances of involved mental representations involved : space-centered neglect (egocentric) and object-centered neglect (allocentric).
Gainotti's drawing copying test | Immediately following first session of occupational therapy.
  Informs us on two kinds of peri-personal neglect referring to distinct disturbances of involved mental representations involved : space-centered neglect (egocentric) and object-centered neglect (allocentric).
Gainotti's drawing copying test | after the first week of protocol
  Informs us on two kinds of peri-personal neglect referring to distinct disturbances of involved mental representations involved : space-centered neglect (egocentric) and object-centered neglect (allocentric).
Gainotti's drawing copying test | After the third week of protocol
  Informs us on two kinds of peri-personal neglect referring to distinct disturbances of involved mental representations involved : space-centered neglect (egocentric) and object-centered neglect (allocentric).
Gainotti's drawing copying test | 3 weeks after the last session of intervention
  Informs us on two kinds of peri-personal neglect referring to distinct disturbances of involved mental representations involved : space-centered neglect (egocentric) and object-centered neglect (allocentric).
The Map of France test | Immediately following first session of occupational therapy.
  The number of cities mentioned will be counted on either side of a median line drawn vertically through the center of France. A mental evocation score will be calculated as the ratio of the number of cities on each side of this axis (left/right). The higher the score, the better the performance.
The Map of France test | After the first experimental session
  The number of cities mentioned will be counted on either side of a median line drawn vertically through the center of France. A mental evocation score will be calculated as the ratio of the number of cities on each side of this axis (left/right). The higher the score, the better the performance.
The Map of France test | After the first week of protocol
  The number of cities mentioned will be counted on either side of a median line drawn vertically through the center of France. A mental evocation score will be calculated as the ratio of the number of cities on each side of this axis (left/right). The higher the score, the better the performance.
The Map of France test | After the third week of protocol
  The number of cities mentioned will be counted on either side of a median line drawn vertically through the center of France. A mental evocation score will be calculated as the ratio of the number of cities on each side of this axis (left/right). The higher the score, the better the performance.
The Map of France test | 3 weeks after the last session of intervention
  The number of cities mentioned will be counted on either side of a median line drawn vertically through the center of France. A mental evocation score will be calculated as the ratio of the number of cities on each side of this axis (left/right). The higher the score, the better the performance.
The Subjective Straight-Ahead test | At the end of the first week of inclusion
  Its investigates the accuracy of egocentric perception. EThe egocentric perception will be expressed as the mean error of 20 successive trials, after measuring for each trial the angular difference between the measured angles of the hand pointed towards SSA direction and the objective straight-ahead direction of the patient's body. A higher score indicates a less accurate egocentric perception.
The Subjective Straight-Ahead test | Immediately following first session of occupational therapy.
  Its investigates the accuracy of egocentric perception. EThe egocentric perception will be expressed as the mean error of 20 successive trials, after measuring for each trial the angular difference between the measured angles of the hand pointed towards SSA direction and the objective straight-ahead direction of the patient's body. A higher score indicates a less accurate egocentric perception.
The Subjective Straight-Ahead test | After the first week of protocol
  Its investigates the accuracy of egocentric perception. EThe egocentric perception will be expressed as the mean error of 20 successive trials, after measuring for each trial the angular difference between the measured angles of the hand pointed towards SSA direction and the objective straight-ahead direction of the patient's body. A higher score indicates a less accurate egocentric perception.
The Subjective Straight-Ahead test | After the third week of protocol
  Its investigates the accuracy of egocentric perception. EThe egocentric perception will be expressed as the mean error of 20 successive trials, after measuring for each trial the angular difference between the measured angles of the hand pointed towards SSA direction and the objective straight-ahead direction of the patient's body. A higher score indicates a less accurate egocentric perception.
The Subjective Straight-Ahead test | 3 weeks after the last session of intervention
  Its investigates the accuracy of egocentric perception. EThe egocentric perception will be expressed as the mean error of 20 successive trials, after measuring for each trial the angular difference between the measured angles of the hand pointed towards SSA direction and the objective straight-ahead direction of the patient's body. A higher score indicates a less accurate egocentric perception.
The Wheelchair navigation test | At the end of the first week of inclusion
  Investigating spatial navigation skills and extra-personal neglect. The ride will be carried out once in each direction (A-B and B-A) to balance the number of obstacles and turns to the left and right. The time taken to finish the course will be measured and the number of bumps counted. Navigation quality will also be observed qualitatively (obstacle avoidance, goal strategy, perseverations).
The Wheelchair navigation test | Immediately following first session of occupational therapy.
  Investigating spatial navigation skills and extra-personal neglect. The ride will be carried out once in each direction (A-B and B-A) to balance the number of obstacles and turns to the left and right. The time taken to finish the course will be measured and the number of bumps counted. Navigation quality will also be observed qualitatively (obstacle avoidance, goal strategy, perseverations).
The Wheelchair navigation test | After the first week of protocol
  Investigating spatial navigation skills and extra-personal neglect. The ride will be carried out once in each direction (A-B and B-A) to balance the number of obstacles and turns to the left and right. The time taken to finish the course will be measured and the number of bumps counted. Navigation quality will also be observed qualitatively (obstacle avoidance, goal strategy, perseverations).
The Wheelchair navigation test | After the third week of protocol
  Investigating spatial navigation skills and extra-personal neglect. The ride will be carried out once in each direction (A-B and B-A) to balance the number of obstacles and turns to the left and right. The time taken to finish the course will be measured and the number of bumps counted. Navigation quality will also be observed qualitatively (obstacle avoidance, goal strategy, perseverations).
The Wheelchair navigation test | 3 weeks after the last session of intervention
  Investigating spatial navigation skills and extra-personal neglect. The ride will be carried out once in each direction (A-B and B-A) to balance the number of obstacles and turns to the left and right. The time taken to finish the course will be measured and the number of bumps counted. Navigation quality will also be observed qualitatively (obstacle avoidance, goal strategy, perseverations).

CONTACTS AND LOCATIONS:
Overall Officials: Hadrien Ceyte, PhD, HDR, Study Director — Université de Lorraine, DevAH (EA3450), Nancy, France

IPD SHARING:
Plan to Share IPD: No